CLINICAL TRIAL: NCT01430546
Title: Phase IV Study on QoL in Relapsed/Refractory Multiple Myeloma When Treated With Lenalidomide
Brief Title: Non-interventional Study on Time to Response and Quality of Life in Relapsed/Refractory Multiple Myeloma When Treated With Lenalidomide in Second Line
Status: Completed | Type: Observational
Sponsor: Hareth Nahi (Other)
Responsible Party: Sponsor-Investigator, Hareth Nahi, MD, PhD, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Other Study IDs: PI-RV-MM-10-06
Record Dates: First submitted 2011-09-07; First posted 2011-09-08 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Myeloma
Keywords: Relapsed and Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to quantify the burden of treatment in relapsed or refractory multiple myeloma in patients receiving lenalidomide after one prior treatment for myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age
2. Have a confirmed diagnosis of MM
3. Starting lenalidomide treatment for MM (due to relapsed or refractory disease) after one prior treatment.
4. Have personally signed and dated a legally effective written informed consent form prior to admission to the study.
5. Must be willing and able to understand and comply with the study requirements.

Exclusion Criteria:

1. Individuals who have taken any experimental drugs or participated in a clinical trial within 30 days prior to screening.
2. Individuals with significant psychiatric illness or a clinically significant acute/chronic uncontrolled medical condition that might affect their experience of myeloma symptoms or their ability to describe them.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2010-11; Primary Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hareth Nahi, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska Institute, Stockholm, Sweden

REFERENCES:
- [Derived] Lund J, Gruber A, Lauri B, Duru AD, Blimark C, Swedin A, Hansson M, Forsberg K, Ahlberg L, Carlsson C, Waage A, Gimsing P, Vangsted AJ, Frolund U, Holmberg E, Gahrton G, Alici E, Hardling M, Mellqvist UH, Nahi H. Lenalidomide versus lenalidomide + dexamethasone prolonged treatment after second-line lenalidomide + dexamethasone induction in multiple myeloma. Cancer Med. 2018 Jun;7(6):2256-2268. doi: 10.1002/cam4.1422. Epub 2018 Apr 19. PMID 29673108